CLINICAL TRIAL: NCT00206193
Title: Termination of Pregnancy With Mifepristone and Misoprostol Versus Sulprostone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atrium Medical Center (Other)
Other Study IDs: TOP-protocol
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2005-09

CONDITIONS: Abortion, Induced
Keywords: termination of pregnancy
MeSH Terms: interventions — Mifepristone; Misoprostol; sulprostone

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: mifepristone
Drug: misoprostol
Drug: sulprostone

SUMMARY:
The purpose of this study is to determine which medical treatment is the most effective to terminate a pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women by whom a termination of pregnancy is desired.

Exclusion Criteria:

* Women with liver/kidney disease
* Women on long-term use of corticosteroids (> 6 months)
* Cardiovascular problems
* Therapy-resistant diabetic women
* Therapy-resistant asthma/bronchitis
* Thalassemia
* Ulcerative colitis
* Peptic ulcer disease
* Glaucoma
* Porphyria
* Allergic reaction to prostaglandin or mifepristone
* Women with a prior caesarian section or women with contractions at the start of the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: F Roumen, Dr., Study Director — Atrium Medisch Centrum, Heerlen
Locations (1):
- Atrium Medisch Centrum, Heerlen, Limburg, Netherlands